CLINICAL TRIAL: NCT05165355
Title: A Phase II, Single-armed Study to Assess the Efficacy and Safety of Furmonertinib in Patients With Epidermal Growth Factor Receptor Mutation Positive Stage IB-IIA Non-small Cell Lung Carcinoma, Following Complete Tumour Resection.
Brief Title: Adjuvant Targeted-therapy for Patients With Resected High-risk EGFR-mutant Stage IB-IIA Non-small Cell Lung Carcinoma
Acronym: ATHEM
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tongji University (Other)
Responsible Party: Principal Investigator, Jiang Fan, Director of department of thoracic surgery, Tongji University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SGHDOT 21-12
Record Dates: First submitted 2021-12-20; First posted 2021-12-21 (Actual); Last update posted 2022-01-18 (Actual); Status verified 2022-01

CONDITIONS: NSCLC; EGF-R Positive Non-Small Cell Lung Cancer
Keywords: NSCLC; EGFR mutation; adjuvant therapy
MeSH Terms: interventions — aflutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group (Experimental): Furmonertinib (80 mg orally, once daily) for 3 years.
  Interventions: Drug: Furmonertinib

INTERVENTIONS:
Drug: Furmonertinib — Furmonertinib (80 mg orally, once daily) for 3 years.

SUMMARY:
This is a single-armed study designed to evaluate the safety and efficacy of adjuvant targeted-therapy in patients with epidermal growth factor receptor mutation positive stage IB-IIA non-small cell lung carcinoma and high-risk of recurrence following complete tumor resection.

The primary endpoint: 2-year DFS rate; The second endpoint: DFS

ELIGIBILITY:
Inclusion Criteria:

1. Subjects aged ≥18 and ≤75 years old；
2. ECOG performance status score 0-1；
3. Stage ⅠB-ⅡA（according to the 8th Edition of the AJCC Staging system）；
4. Complete surgical resection of the primary NSCLC is mandatory；
5. Histologically confirmed diagnosis of high-risk pathological subtype (micropapillary, solid pattern or spread through air spaces [STAS], etc.);
6. The tumour harbours one of the most common EGFR mutations (19del or L858R) ;
7. Normal organ and bone marrow function measured before the study as defined below:

1) Hemoglobin (HGB)≥90g/L 2) White blood cell count (WBC) is 4.0~10×10^9/L 3) Absolute value of neutrophil (ANC)≥1.5×10^9/L 4) Platelet (PLT) count≥100×109/L 5) Serum total bilirubin (TBIL)≤1.5×ULN 6) AST and/or ALT≤2.5×ULN 7) International normalized ratio（INR）≤1.5 and activated partial thromboplastin time (APTT) is normal 8) Serum creatinine (SCr)≤1.5 × ULN 8. No previous systemic anti-tumor therapy for malignant tumor, such as chemotherapy, radiotherapy or hormonotherapy. No history of other malignancies, subjects with prostate cancer who received hormone therapy and had more than 5 years of DFS were excluded; 9. Subjects have voluntarily participated, signed and dated informed consent.

Exclusion Criteria:

1. Double primary lung cancer or multiple primary lung cancer;
2. Subjects with mental illness;
3. Presence or concomitant hemorrhagic diseases;
4. Pregnancy or lactation;
5. Known or suspected to be allergic to Furmonertinib and / or other components of their preparations.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2021-12-28 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Disease Free Survival (DFS) rate at 2 years | From date of receiving therapy until date of disease recurrence or death (by any cause in the absence of recurrence), up to approximately 4 years. Assessed at 2 years.
  Assess the Efficacy of Adjuvant Furmonertinib as Measured by 2-year Disease Free Survival (DFS) rate.

SECONDARY OUTCOMES:
Disease Free Survival (DFS) | From date of receiving therapy until date of disease recurrence or death (by any cause in the absence of recurrence), up to approximately 4 years.
  Assess the Efficacy of Adjuvant Furmonertinib as Measured by Disease Free Survival (DFS).

CONTACTS AND LOCATIONS:
Overall Officials: Jiang Fan, MD, Principal Investigator — Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Locations (1):
- Shanghai General Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No